CLINICAL TRIAL: NCT04441437
Title: The Efficacy of Dynamic Hand Splint Treatment in Spastic Hemiparetic Patients: A Randomized Controlled Trial
Brief Title: The Efficacy of Dynamic Hand Splint Treatment in Spastic Hemiparetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chu-Hsu Lin, Principal Investigator, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 104-9569A3
Record Dates: First submitted 2020-06-16; First posted 2020-06-22 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Stroke; Brain Injuries
Keywords: spasticity; dynamic hand splint; stroke; traumatic brain injury
MeSH Terms: conditions — Stroke; Brain Injuries; Muscle Spasticity; Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Splint Group (Experimental): 1-hour task-oriented training with wearing a customized dynamic hand splint, totally 15 times in a duration of one month.
  Interventions: Behavioral: Task-oriented training with a dynamic hand splint
- No-Splint Group (Placebo Comparator): 1-hour task-oriented training without wearing a customized dynamic hand splint, totally 15 times in a duration of one month.
  Interventions: Behavioral: Task-oriented training without a dynamic hand splint

INTERVENTIONS:
Behavioral: Task-oriented training with a dynamic hand splint — In addition to conventional rehabilitation programs (therapy-as-usual), the subject in the splint group received 1-hour task-oriented training with wearing a customized dynamic hand splint, totally 15 times in a duration of one month. The content of task-oriented training contained picking cubes from side to side with three-jaw grasp, lifting the cone to the shoulder height with the cylindrical grip and an extended elbow, picking up pegs and inserting it into the hole with palmar pinch, and grasping a soap to simulate wiping the body. Among the four tasks, two were chosen to train the subjects according to the abilities of subjects.
  Arms: Splint Group
Behavioral: Task-oriented training without a dynamic hand splint — In addition to conventional rehabilitation programs (therapy-as-usual), the subject in the no-splint group received 1-hour task-oriented training, totally 15 times in a duration of one month. The content of task-oriented training contained picking cubes from side to side with three-jaw grasp, lifting the cone to the shoulder height with the cylindrical grip and an extended elbow, picking up pegs and inserting it into the hole with palmar pinch, and grasping a soap to simulate wiping the body. Among the four tasks, two were chosen to train the subjects according to the abilities of subjects.
  Arms: No-Splint Group

SUMMARY:
The purpose of this randomized controlled trial was designed to study the efficacy of dynamic hand splinting on spastic hemiparetic patients due to stroke or traumatic brain injury.

DETAILED DESCRIPTION:
Subjects were recruited from both inpatients and outpatients who received rehabilitation programs in the Department of Physical Medicine and Rehabilitation at a regional teaching hospital in Taiwan. The participants were randomly divided into two groups: the splint group and the control group. The subjects in the splint group received 1-hour task-oriented training with wearing a customized dynamic hand splint, totally 15 times in a duration of one month plus conventional rehabilitation programs. The subjects in the control group received the same treatments but without splint used. Evaluations including Modified Ashworth Scale (MAS), active range of motion (AROM), grip strength, Fugl-Meyer Assessment (FMA), Motor Activity Log 30(MAL), and F/M ratio were performed at baseline, post-training, and 2 months later after the intervention finished, and the evaluators were blinded to the grouping of the subjects.

ELIGIBILITY:
Inclusion Criteria:

* an age of 20 to 85 years
* the duration of stroke or brain injury more than 6 months
* unilateral hemiparesis with intact sound side limbs function
* the Brunnstrom's stage of both arm and hand ≥ III
* able to follow instructions, wear a dynamic hand splint and perform therapeutic activities
* wrist spasticity with a Modified Ashworth Scale score 1-3
* willing to provide the written informed consent.

Exclusion Criteria:

* patients with apraxia
* cognitive impairment with a Mini-Mental State Examination (MMSE) score < 25
* any fixed contracture of the affected wrist or fingers
* a history of peripheral nerve injury, other severe neuromuscular disease or musculoskeletal deformity change in the affected side upper extremity
* a history of alcohol or phenol injection to the affected side upper extremity
* Botulinum toxin injection to the affected side upper extremity for the treatment of spasticity within 4 months before the study
* surgical treatment for spasticity to the affected side upper extremity
* active infection
* obvious atrophy of muscles in the affected side upper extremity
* bilateral upper extremities weakness
* any dermatosis or open wounds in the affected upper extremity or an allergy to the splint.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-11-04 (Actual); Primary Completion 2019-03-22 (Actual); Study Completion 2019-03-22 (Actual)

PRIMARY OUTCOMES:
Modified Ashworth Scale (MAS) | Performed at baseline
  A participant was made in sitting position with the palm of the affected side placed at the edge of table. Then his or her 2nd to 5th fingers was moved by the examiner from maximum possible flexion to maximum possible extension over a duration of about one second. All of the four fingers were done at once. The participant's wrist and elbow were then also tested in the same manner. The lowest score was zero and the highest score was 415. For statistical purposes, the MAS score '1+' is considered as 2, '2' as 3, and so on until 5.
Post-training Change of Modified Ashworth Scale (MAS) | Change from baseline at average 30 days
  A participant was made in sitting position with the palm of the affected side placed at the edge of table. Then his or her 2nd to 5th fingers was moved by the examiner from maximum possible flexion to maximum possible extension over a duration of about one second. All of the four fingers were done at once. The participant's wrist and elbow were then also tested in the same manner. The lowest score was zero and the highest score was 415. For statistical purposes, the MAS score '1+' is considered as 2, '2' as 3, and so on until 5.
3-Month Follow-up Change of Modified Ashworth Scale (MAS) | Change from baseline at average 90 days
  A participant was made in sitting position with the palm of the affected side placed at the edge of table. Then his or her 2nd to 5th fingers was moved by the examiner from maximum possible flexion to maximum possible extension over a duration of about one second. All of the four fingers were done at once. The participant's wrist and elbow were then also tested in the same manner. The lowest score was zero and the highest score was 415. For statistical purposes, the MAS score '1+' is considered as 2, '2' as 3, and so on until 5.
Active range of motion (AROM) | Performed at baseline
  A participant in sitting position with the palm of the affected side placed at the edge of table was instructed to actively move his or her fingers and wrists as much as possible. Then the AROM of the index finger and wrist were measured by a goniometer.
Post-training Change of Active range of motion (AROM) | Change from baseline at average 30 days
  A participant in sitting position with the palm of the affected side placed at the edge of table was instructed to actively move his or her fingers and wrists as much as possible. Then the AROM of the index finger and wrist were measured by a goniometer.
3-Month Follow-up Change of Active range of motion (AROM) | Change from baseline at average 90 days
  A participant in sitting position with the palm of the affected side placed at the edge of table was instructed to actively move his or her fingers and wrists as much as possible. Then the AROM of the index finger and wrist were measured by a goniometer.
Grip strength | Performed at baseline
  For the grip strength measurement, a participant in sitting position was instructed to squeeze a dynamometer with the unaffected hand as hard as he or she can for about 3 seconds. Then the hand of affected side was tested in the same manner. Three consecutive measurements with a 3-minute interval were performed for each hand and the arithmetic mean value of the 3 trials was used for statistical analysis.
Post-training Change of Grip strength | Change from baseline at average 30 days
  For the grip strength measurement, a participant in sitting position was instructed to squeeze a dynamometer with the unaffected hand as hard as he or she can for about 3 seconds. Then the hand of affected side was tested in the same manner. Three consecutive measurements with a 3-minute interval were performed for each hand and the arithmetic mean value of the 3 trials was used for statistical analysis.
3-Month Follow-up Change of Grip strength | Change from baseline at average 90 days
  For the grip strength measurement, a participant in sitting position was instructed to squeeze a dynamometer with the unaffected hand as hard as he or she can for about 3 seconds. Then the hand of affected side was tested in the same manner. Three consecutive measurements with a 3-minute interval were performed for each hand and the arithmetic mean value of the 3 trials was used for statistical analysis.
Motor Activity Log 30(MAL) | Performed at baseline
  Using the standardized questions from the upper-extremity MAL, a participant was rated how much (Amount of Use scale, MAL-AOU) and how well (Quality of Movement scale, MAL-QOM) he or she used the upper limb of affected side to accomplish each functional activity during the past week. Both scales were anchored at 6 points (AOU scale: 0 = not used, 5 = the same as before stroke or brain injury; QOM scale: 0 = not used, 5 = normal).17, 18 A mean MAL score is the mean of all item scores.
Post-training Change of Motor Activity Log 30(MAL) | Change from baseline at average 30 days
  Using the standardized questions from the upper-extremity MAL, a participant was rated how much (Amount of Use scale, MAL-AOU) and how well (Quality of Movement scale, MAL-QOM) he or she used the upper limb of affected side to accomplish each functional activity during the past week. Both scales were anchored at 6 points (AOU scale: 0 = not used, 5 = the same as before stroke or brain injury; QOM scale: 0 = not used, 5 = normal).17, 18 A mean MAL score is the mean of all item scores.
3-Month Follow-up Change of Motor Activity Log 30(MAL) | Change from baseline at average 90 days
  Using the standardized questions from the upper-extremity MAL, a participant was rated how much (Amount of Use scale, MAL-AOU) and how well (Quality of Movement scale, MAL-QOM) he or she used the upper limb of affected side to accomplish each functional activity during the past week. Both scales were anchored at 6 points (AOU scale: 0 = not used, 5 = the same as before stroke or brain injury; QOM scale: 0 = not used, 5 = normal).17, 18 A mean MAL score is the mean of all item scores.
Fugl-Meyer Assessment (FMA) | Performed at baseline
  For the Fugl-Meyer Upper Extremity Assessment (FMA), a 3-graded scale with 0 as minimum and 2 as maximum was applied for grading of sensorimotor function.19 The testing procedure was conducted in a standardized manner according to the written instructions originally published and some additional general guidelines.20, 21 For motor function assessment, the Fugl-Meyer Assessment for upper extremity (FMA-UE) was used. Clear and precise instructions were given to a seated participant for each movement. The unaffected side simulated first and then the affected side was evaluated. Each activity was repeated 3 times and the highest score was recorded. The maximum total score was 66. For sensory function assessment, the Modified Fugl-Meyer sensory assessment (FMA-sensory) was used. This included tests of the light touch, temperature, tactile localization and position sensation of the upper arm, forearm, hand, thigh, calf and foot of the affected side. The maximum total score was 44.
Post-training Change of Fugl-Meyer Assessment (FMA) | Change from baseline at average 30 days
  For the Fugl-Meyer Upper Extremity Assessment (FMA), a 3-graded scale with 0 as minimum and 2 as maximum was applied for grading of sensorimotor function.19 The testing procedure was conducted in a standardized manner according to the written instructions originally published and some additional general guidelines.20, 21 For motor function assessment, the Fugl-Meyer Assessment for upper extremity (FMA-UE) was used. Clear and precise instructions were given to a seated participant for each movement. The unaffected side simulated first and then the affected side was evaluated. Each activity was repeated 3 times and the highest score was recorded. The maximum total score was 66. For sensory function assessment, the Modified Fugl-Meyer sensory assessment (FMA-sensory) was used. This included tests of the light touch, temperature, tactile localization and position sensation of the upper arm, forearm, hand, thigh, calf and foot of the affected side. The maximum total score was 44.
3-Month Follow-up Change of Fugl-Meyer Assessment (FMA) | Change from baseline at average 90 days
  For the Fugl-Meyer Upper Extremity Assessment (FMA), a 3-graded scale with 0 as minimum and 2 as maximum was applied for grading of sensorimotor function.19 The testing procedure was conducted in a standardized manner according to the written instructions originally published and some additional general guidelines.20, 21 For motor function assessment, the Fugl-Meyer Assessment for upper extremity (FMA-UE) was used. Clear and precise instructions were given to a seated participant for each movement. The unaffected side simulated first and then the affected side was evaluated. Each activity was repeated 3 times and the highest score was recorded. The maximum total score was 66. For sensory function assessment, the Modified Fugl-Meyer sensory assessment (FMA-sensory) was used. This included tests of the light touch, temperature, tactile localization and position sensation of the upper arm, forearm, hand, thigh, calf and foot of the affected side. The maximum total score was 44.
F/M ratio of ulnar nerve | Performed at baseline
  An electrophysiological examination was performed with an active recording surface electrode (G1) placed over the belly of the abductor digiti minimi of the affected side, a reference electrode (G2) placed on the phalanx of the little finger, and a ground electrode placed on the back of the hand between the stimulating and recording electrodes. Supra-maximal stimulations at the wrist 8 cm away from G1 was performed to obtain the compound muscle action potential (CMAP) and F wave of the ADM muscle with the cathode distal and proximal to the anode, respectively. The stimulation was given less than 1 Hz to avoid influences from the previous stimulus. The ratio of amplitude of the mean and the maximal F-wave to the CMAP (F/M ratio) were then calculated.
Post-training Change of F/M ratio of ulnar nerve | Change from baseline at average 30 days
  An electrophysiological examination was performed with an active recording surface electrode (G1) placed over the belly of the abductor digiti minimi of the affected side, a reference electrode (G2) placed on the phalanx of the little finger, and a ground electrode placed on the back of the hand between the stimulating and recording electrodes. Supra-maximal stimulations at the wrist 8 cm away from G1 was performed to obtain the compound muscle action potential (CMAP) and F wave of the ADM muscle with the cathode distal and proximal to the anode, respectively. The stimulation was given less than 1 Hz to avoid influences from the previous stimulus. The ratio of amplitude of the mean and the maximal F-wave to the CMAP (F/M ratio) were then calculated.
3-Month Follow-up Change of F/M ratio of ulnar nerve | Change from baseline at average 90 days
  An electrophysiological examination was performed with an active recording surface electrode (G1) placed over the belly of the abductor digiti minimi of the affected side, a reference electrode (G2) placed on the phalanx of the little finger, and a ground electrode placed on the back of the hand between the stimulating and recording electrodes. Supra-maximal stimulations at the wrist 8 cm away from G1 was performed to obtain the compound muscle action potential (CMAP) and F wave of the ADM muscle with the cathode distal and proximal to the anode, respectively. The stimulation was given less than 1 Hz to avoid influences from the previous stimulus. The ratio of amplitude of the mean and the maximal F-wave to the CMAP (F/M ratio) were then calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Chu-Hsu Lin, MD, Principal Investigator — Chang Gung Memorial Hospital

IPD SHARING:
Plan to Share IPD: No